CLINICAL TRIAL: NCT01079013
Title: Phase II Trial of Fludarabine Combined With Intravenous Treosulfan and Allogeneic Hematopoietic Stem-cell Transplantation in Patients With Lymphatic Malignancies
Brief Title: Treosulfan-based Conditioning for Allogeneic Stem-cell Transplantation (SCT) in Lymphoid Malignancies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-09-7425-AN-CTIL
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Non Hodgkin Lymphoma; Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — treosulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treosulfan (Experimental)
  Interventions: Drug: treosulfan

INTERVENTIONS:
Drug: treosulfan — 12 g/m2 x 3 days

SUMMARY:
The study hypotheses is that the introduction of dose escalated treosulfan, in substitution to busulfan or melphalan, will reduce toxicity after allogeneic transplantation while improving disease eradication in patients with lymphoid malignancies not eligible for standard transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age less than physiologic 68 years.
2. Patients with NHL and HL with an indication for allogeneic transplantation as follows:

   * Aggressive lymphoma and Hodgkin lymphoma; relapse after autologous transplants
   * Follicular lymphoma; failure of at least one prior regimen
3. Disease must be at chemo-sensitive or stable status to prior therapy before transplant.
4. Patients must have an HLA matched related or unrelated donor willing to donate either peripheral blood stem cells or bone marrow. Matching is based on high-resolution class I (HLA-A, -B, -C) and class II (HLA-DRB1, -DQB1) typing. The goal is to transplant > 3 x 106 CD34+ cells per kg body weight of the recipient
5. Patients must sign written informed consent
6. Adequate birth control in fertile patients

Exclusion Criteria:

1. Overt progressive disease prior to transplantation.
2. Bilirubin > 3.0 mg/dl, transaminases > 3 times upper normal limit
3. Creatinine > 2.0 mg/dl
4. ECOG-Performance status > 2
5. Uncontrolled infection
6. Pregnancy or lactation
7. Abnormal lung diffusion capacity (DLCO < 40% predicted)
8. Severe cardiovascular disease
9. CNS disease involvement
10. Pleural effusion or ascites > 1 liter
11. Known hypersensitivity to fludarabine or treosulfan
12. Psychiatric conditions/disease that impair the ability to give informed consent or to adequately co-operate

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-03; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 2 years after transplantation

SECONDARY OUTCOMES:
treatment-related mortality | 2 year after transplantation
GVHD | 2 year after transplantation
relapse | 2 year after transplantation
overall survival | 2 year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Nagler, MD, Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Tel Litwinsky, Tel-Hashomer, Israel